CLINICAL TRIAL: NCT01209936
Title: Pilot Study for the Validation of the BC3 Bioelectrical Impedance Hydration Factor
Brief Title: Hydration Factor Study for the Stayhealthy BC3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Todd Schroeder, Associate Professor, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Stayhealthy 02
Record Dates: First submitted 2010-09-24; First posted 2010-09-27 (Estimated); Results first posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Body Composition
Keywords: Body Fat; Total body water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- deuterium oxide and BC3 (Experimental): Testing of total body water on the BC3 compared to total body water measured by deuterium oxide.
  Interventions: Device: D2O

INTERVENTIONS:
Device: D2O — All participants received deuterium oxide (D2O) and testing with the BC3 for the measurement of total body water.
  Other Names: Stayhealthy BC3 Body Composition Analyzer

SUMMARY:
This was a pilot study to validate the BC3 hydration factor which will be important for determining how well this value represents hydration status compared to assessment of total body water by D20.

DETAILED DESCRIPTION:
The BC3 body composition analyzer is manufactured by Stayhealthy. It is a handheld, noninvasive bioelectrical impedance device. When held, the BC3 sends an electrical impulse through the body to determine body fat, lean mass, and total body hydration. Bio-impedance devices measure the change in electrical resistance in body tissues by using a detectable electrical signal that passes through the body. The method is based on the principle that lean body mass contains virtually all the water and conducting electrolytes in the body and provides a good electrical pathway. In contrast, fat or fat-containing tissues produce a poor electrical pathway. By inducing a low-energy, high-frequency signal, a measurement of the baseline resistance to flow of electrical current can be assessed. The resistance measurement relates directly to the volume of the conductor. Through repeated measurements and identifying other parameters (i.e. gender, weight, age and height) proprietary equations were developed that determine total body water, lean mass, and % body fat.

The purpose of this study is to validate the calculated hydration factor produced by the BC3 bioelectrical impedance device. If this value is valid and comparable to the gold standard (D20) then this hydration factor will offer a very quick and inexpensive method to determine total body hydration status using a hand-held bioelectrical impedance device.

ELIGIBILITY:
Inclusion Criteria:

• Men and women 18-80 years of age

Exclusion Criteria:

* Acute illness (infection, recent surgery, trauma).
* Pregnancy
* Pacemaker or defibrillator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2009-09; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward T Schroeder, PhD, Principal Investigator — University of Southern California
Locations (1):
- USC Clinical Exercise Research Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Adults: All adults underwent a 10-15 minute total body DXA Scan. All adults used the Stayhealthy body composition analyzer BC3 for BIA to measure body composition.
  All participants received deuterium oxide (D2O) and testing with the BC3 for the measurement of total body water.
- Children: All children were measured using Hydrostatic Weighing (HW) to assess body composition, a DEXA was not used to avoid unnecessary radiation exposure. HW was measured by placing the participants in a chair suspended from spring-loaded scale inside a plexiglass tank. Weight was averaged among 3 trials, that fell within 100g of each other. Density was adjusted for residual volume using an estimated volume of 115 mL. % body fat was calculated using Lohman's equations to adjust for age and sex.
  All children used the Stayhealthy body composition analyzer BC3 for BIA to measure body composition.
  All participants received deuterium oxide (D2O) and testing with the BC3 for the measurement of total body water.
Period: Overall Study
Arm/Group | Adults | Children
Started | 245 | 115
Completed | 245 | 115
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Children: All children were measured using Hydrostatic Weighing to assess body composition. All children used the Stayhealthy body composition analyzer BC3 for BIA to measure body composition.
  All participants received deuterium oxide (D2O) and testing with the BC3 for the
- Total: Total of all reporting groups
Arm/Group | Adults | Children | Total
Number analyzed (Participants) | 245 | 115 | 360
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.4 (16.75) | 14.9 (1.7) | 30.15 (9.225)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 64 | 192
  Male | 117 | 51 | 168
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 245 | 115 | 360

OUTCOME MEASURES:

1. Primary Outcome: Estimated Body Fat % for Children Aged 10-17 Years Old
Description: Stayhealthy BC3 was analyzed against hydrostatic weighing for children aged 10-17 years old
Time Frame: One time point (only one day visit)
Measure: Mean (Standard Deviation); unit: Percent body fat
Groups:
- Estimated Body Fat % From BC3 for Children Aged 10-17 Years Old: The body fat percentage as measured by the Stayhealthy body composition analyzer BC3
Arm/Group | Estimated Body Fat % From BC3 for Children Aged 10-17 Years Old
Number analyzed (Participants) | 115
Percent body fat
  BC3 | 18.4 (8.4)
  Hydrostatic Weighing | 18.8 (8.3)
Statistical Analysis 1: Comparison: Estimated Body Fat % From BC3 for Children Aged 10-17 Years Old; Test type: Superiority; p = 0.87, t-test, 2 sided

2. Primary Outcome: Percent Body Fat in Women Aged 18-80 Years Old
Description: Body fat percentage was measured via Stayhealthy BC3 as well as a full body DXA
Time Frame: One time point (only one day visit)
Measure: Mean (Standard Deviation); unit: Percent body fat
Groups:
- Estimated Percent Body Fat for Women Aged 18-80 Years Old: Body fat percentage from the stayhealthy BC3 was and a full body DXA was used to estimate body fat percentage.
Arm/Group | Estimated Percent Body Fat for Women Aged 18-80 Years Old
Number analyzed (Participants) | 128
Percent body fat
  BC3 | 32.8 (9.1)
  DXA | 33.4 (9.6)
Statistical Analysis 1: Comparison: Estimated Percent Body Fat for Women Aged 18-80 Years Old; Test type: Superiority; p = 0.17, t-test, 2 sided

3. Primary Outcome: Estimated Percent Body Fat for Men Aged 18-80
Description: The body fat percentage as estimated from BC3 and as calculated by a full body DXA.
Time Frame: One time point (only one day visit)
Measure: Mean (Standard Deviation); unit: Percent body fat
Groups:
- Estimated Body Fat Percentage for Men Aged 18-80: Stayhealthy BC3 body fat percentage and as calculated by DXA.
Arm/Group | Estimated Body Fat Percentage for Men Aged 18-80
Number analyzed (Participants) | 117
Percent body fat
  BC3 | 20.3 (5.3)
  DXA | 20.4 (5.6)
Statistical Analysis 1: Comparison: Estimated Body Fat Percentage for Men Aged 18-80; Test type: Superiority; p = 0.55, t-test, 2 sided

ADVERSE EVENTS:
Groups:
- Deuterium Oxide and BC3 Adult; Deuterium Oxide and BC3 Children: Testing of total body water on the BC3 compared to total body water measured by deuterium oxide.
  D2O: All participants received deuterium oxide (D2O) and testing with the BC3 for the measurement of total body water.
Arm/Group | Deuterium Oxide and BC3 Adult | Deuterium Oxide and BC3 Children
Serious Adverse Events (participants affected / at risk) | 0/245 | 0/117
Other Adverse Events (participants affected / at risk) | 0/245 | 0/117

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No